CLINICAL TRIAL: NCT01471717
Title: A Phase Ib, Single-Center, Randomized, Two-Sequence, Placebocontrolled, Drug-Drug Interaction Study to Evaluate the Pharmacokinetics and Safety of INX-08189 Administered With VictrelisTM in Healthy Subjects
Brief Title: Study to Evaluate the Pharmacokinetics and Safety of INX-08189 Administered With VictrelisTM in Healthy Subjects
Acronym: INX-189-004
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: AI472-004; INX-189-004 (Other: INX-189-004)
Record Dates: First submitted 2011-11-03; First posted 2011-11-16 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: PK; pharmacokinetics; INX08189; Victrelis; Inhibitex
MeSH Terms: interventions — BMS-986094; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- C 1:INX-08189 50 mg qd X 5 days (Experimental): Cohort 1: Subjects will begin administration of INX-08189 50 mg every day (QD) on Study Day 0. Dosing will occur each morning for 5 days after a fast of at least 8 hours prior to each dose on Study Days 0 through 4. INX-08189 will be administered with water, and subjects will remain fasting for 2 hours following each dose.
  Interventions: Drug: INX-08189 50 mg QD X 5 days
- C1: INX-08189 / Victrelis 800 mg TID X 3 days (Active Comparator): Cohort 1:INX-08189 50 mg QD will be administered concurrently with Victrelis 800 mg three times a day (TID) for 3 additional days
  Interventions: Drug: INX-08189 / Victrelis 800 mg TID X three days
- C2: Victrelis 800 mg TID x 3 days (Active Comparator): Cohort 2: Subjects will begin administration of Victrelis 800 mg three times a day (TID) on the morning of Study Day 0. Victrelis will be administered with water and food with doses at least 7 hours apart. Victrelis 800 mg TID will be administered for a total of 3 days
  Interventions: Drug: Victrelis 800 mg TID x 3 days
- C 2:Victrelis 800 mg TID with INX-08189 50 mg QD (Active Comparator): Cohort 2: Victrelis 800 mg TID will be administered concurrently with INX-08189 50 mg QD for 5 additional days
  Interventions: Drug: Victrelis 800 mg TID with INX-08189 50 mg QD
- C1: Placebo with Victrelis 800 mg (Placebo Comparator): Cohort 1: Placebo QD will be administered concurrently with Victrelis 800 mg TID for 3 additional days
  Interventions: Drug: Placebo with Victrelis 800 mg
- C 2: Victrelis 800 mg with Placebo (Placebo Comparator): Cohort 2: Victrelis 800 mg TID will be administered concurrently with Placebo QD for 5 additional days
  Interventions: Drug: Cohort 2: Victrelis 800 mg with Placebo

INTERVENTIONS:
Drug: INX-08189 50 mg QD X 5 days — Cohort 1: Subjects will begin administration of INX-08189 50 mg QD on Study Day 0. Dosing will occur each morning for 5 days after a fast of at least 8 hours prior to each dose on Study Days 0 through 4. INX-08189 will be administered with water, and subjects will remain fasting for 2 hours following each dose.
  Arms: C 1:INX-08189 50 mg qd X 5 days
Drug: INX-08189 / Victrelis 800 mg TID X three days — Cohort 1: INX-08189 50 mg QD will be administered concurrently with Victrelis 800 mg TID for 3 additional days (Study Days 5 through 7)
  Arms: C1: INX-08189 / Victrelis 800 mg TID X 3 days
Drug: Victrelis 800 mg TID x 3 days — In Cohort 2, subjects will begin administration of Victrelis 800 mg TID on the morning of Study Day 0. Victrelis will be administered with water and food with doses at least 7 hours apart. Victrelis 800 mg TID will be administered for a total of 3 days (Study Days 0 through 2).
  Arms: C2: Victrelis 800 mg TID x 3 days
Drug: Victrelis 800 mg TID with INX-08189 50 mg QD — Victrelis 800 mg TID will be administered concurrently with INX-08189 50 mg QD for 5 additional days (Study Days 3 through 7).
  Arms: C 2:Victrelis 800 mg TID with INX-08189 50 mg QD
Drug: Placebo with Victrelis 800 mg — During combination dosing with INX-08189 and Victrelis, each morning dose will start with INX-08189 or placebo after at least an 8 hour fast, followed by a 2 hour fast with the first Victrelis dose of the day then administered with food.
  Arms: C1: Placebo with Victrelis 800 mg
Drug: Cohort 2: Victrelis 800 mg with Placebo — During combination dosing with INX-08189 and Victrelis, each morning dose will start with INX-08189 or placebo after at least an 8 hour fast, followed by a 2 hour fast with the first Victrelis dose of the day then administered with food.
  Arms: C 2: Victrelis 800 mg with Placebo

SUMMARY:
This study is designed to evaluate the potential for a pharmacokinetic drug-drug interaction between INX-08189 and Victrelis, a Direct Acting Antiviral (DAA).

DETAILED DESCRIPTION:
This is a single-center, randomized, placebo-controlled study in thirty-two 18 to 55 year old, male and female, healthy adult volunteers.

Primary Objectives:

Pharmacokinetic

* To characterize the pharmacokinetic (PK) profile of INX-08189 and INX-08032 when INX-08189 is dosed alone as compared to when dosed in combination with Victrelis
* To characterize the PK profile of Victrelis when dosed alone as compared to when dosed in combination with INX-08189

Safety

- To evaluate the safety of INX-08189 and Victrelis when dosed alone and when dosed in combination

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria at the Screening Visit (Visit1), in order to be eligible for study drug administration at Study Day 0 (Visit 3):

1. Must be a healthy male or female between 18 and 55 years of age (inclusive) with body mass index (BMI) between 18 and 30 kg/m2 (inclusive), and weigh ≥ 50 kg at the time of signing the informed consent;
2. Capable of giving written informed consent that includes compliance with the requirements and restrictions listed in the consent form. Signed informed consent must be on file prior to screening procedures;
3. Subject is able to understand and comply with the protocol requirements, instructions and restrictions;
4. Must be a non-tobacco user for at least 3 months prior to selection;
5. Healthy on the basis of physical examination, medical history, vital signs, electrocardiogram and clinical laboratory tests at screening;
6. Women must be postmenopausal for at least 2 years or be surgically sterile with complete hysterectomy or bilateral oophorectomy, and not be pregnant nor breastfeeding;
7. Male subjects, who are not surgically sterile with vasectomy, must agree to use a double barrier method of birth control, such as, a condom plus spermicidal agent (foam/gel/film/cream/suppository). This criterion must be followed from the time of the first dose of study medication until 30 days after the last dose of medication. Male subjects cannot donate sperm during the study and for 3 months after receiving the last dose of the study drug.

Exclusion Criteria:

Subjects must NOT meet the following criteria at the Screening Visit (Visit1), in order to be eligible for study drug administration at Study Day 0 (Visit 3):

1. Infection with Hepatitis A, B or C Virus;
2. Infection with the Human Immunodeficiency Virus (HIV);
3. History of or any current medical condition which could impact the safety of the participant in the study;
4. Current active or underlying gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease;
5. Clinically significant abnormalities on centrally read ECG;
6. Currently significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability;
7. Safety laboratory abnormalities at screening which are clinically significant, or absolute neutrophil count of < 1800 cells/mm3, or platelet count < 130,000 cells/mm3, or hemoglobin < 12 g/dl for women and < 13 g/dl for men;
8. Women of child bearing potential;
9. Pregnant or breastfeeding;
10. Current abuse of alcohol or illicit drugs, or history of alcohol or illicit drug abuse within the preceding two years;
11. A positive urine drug test at screening;
12. Consumption of more than 2 units of alcoholic beverages per day or more than 14 units per week (1 unit of alcohol equals 1 glass of beer, 1 glass of wine, 25ml shot of 40% spirit), consumption of alcohol 72 hours before or after study medication intake, consumption of an average of more than five 240 ml servings of coffee or other caffeinated beverages per day;
13. Use of chronic prescription medications within 3 months, acute prescription medications within 14 days, or systemic over-the-counter (OTC) medications, including vitamins, within 7 days of starting the study;
14. Received an investigational drug or vaccine within 30 days or 5 half lives, whichever is longer, from the receipt of a small molecule or 90 days or 5 half lives, whichever is longer, from the receipt of a large biological molecule prior to Study Day 0, or used an investigational medical device within 30 days prior to Study Day 0, or having participated previously in a study with INX-08189.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
PK parameters of INX-08189, INX-08032, and Victrelis when dosed alone and in combination | INX-08189: C1: Days 4 & 7; C2: Day 7 pre-dose & 15, 30, & 45 minutes, & 1, 2, 3, 4, 6, 8, 10, 12, 16, & 24 hours after dosing. Victrelis: C2: Days 2 & 7; C1: Day 7 pre-dose & 0.5, 1, 2, 3, 4, 6, & 8 hours after AM dose. Up to 72 hours after last dose.
  PK parameters of INX-08189, INX-08032, and Victrelis when dosed alone and in combination: maximum observed plasma concentration (Cmax), time at which Cmax is observed (Tmax), plasma concentration at the end of dosing interval (Ctau), area under the plasma concentration-time curve from time 0 to the end of dosing interval (AUC0-tau), elimination half-life (t1/2), apparent oral clearance (CL/F), and apparent oral volume of distribution (Vz/F), as applicable
Safety parameters, including adverse event, concurrent medication, clinical laboratory, ECG, PE, and VS assessments | Study Day 1 to 8, and Study Day 14
  Safety will be monitored by PEs, VS, clinical laboratory tests (including blood chemistry, CBC with differential, Troponin I, creatinine phosphokinase, and urinalysis), ECGs, and AE assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Campaneria, MD, Study Director
Locations (1):
- Prism Research, LLC, Saint Paul, Minnesota, United States